CLINICAL TRIAL: NCT05553548
Title: Alveolar Ridge Changes With Biologically Oriented Alveolar Ridge Preservation (BARP) After Tooth Extraction : A Randomized Clinical Trial
Brief Title: Alveolar Ridge Changes With Biologically Oriented Alveolar Ridge Preservation (BARP) After Tooth Extraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nevein Mohammed Osama Al-Gammal, Assisstant lecturer In periodontology department Future university in Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8722
Record Dates: First submitted 2022-09-18; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Alveolar Ridge Preservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biologically oriented alveolar ridge preservation (BARP) group (Experimental): for alveolar ridge preservation using demineralized bovine bone graft layer in the most coronal part of the extracted tooth socket
  Interventions: Procedure: biologically oriented alveolar ridge preservation
- bone graft (entire apico-coronal extension) (Active Comparator): alveolar ridge preservation using demineralized bovine bone graft on the entire apico-coronal extension.
  Interventions: Procedure: xenogenic bone graft in entire (apico-coronal) extension

INTERVENTIONS:
Procedure: biologically oriented alveolar ridge preservation — xenogenic bone graft placed in coronal part of the non molar socket ,, collagen plug placed in appical part of socket and as socket seal
  Arms: biologically oriented alveolar ridge preservation (BARP) group
Procedure: xenogenic bone graft in entire (apico-coronal) extension — xenogenic bone graft placed in the entire apico coronal extension and sealed with collagen plug
  Arms: bone graft (entire apico-coronal extension)

SUMMARY:
After tooth extraction, the alveolar process undergoes substantial horizontal and vertical resorption specifically in non-molar sites, where horizontal, vertical mid- facial, and mid-lingual ridge reduction could occur . These dimensional changes are clinically relevant, as they may affect dental implant placement and compromise soft tissue aesthetics.

Alveolar ridge preservation (ARP) is based on the application of a bone replacement graft into the extraction socket & collagen membrane/plug. Recent systematic reviews have shown that ARP may limit bone resorption to about 50% of what is normally observed in case of unassisted healing . This finding indicates that ARP is effective; but at the same time, it underlines the potential for improvement.

DETAILED DESCRIPTION:
In ARP procedures based on socket grafting, the use of a bone replacement graft would prevent up to a 30% of volume reduction in the coronal third. Whereas it has limited effect in the remaining middle-apical thirds . Since grafting of the alveolus often results in the persistence of residual graft particles embedded into the newly formed bone with a delay in the rate of bone deposition and mineralization the need to extend the grafting procedure apical to the coronal third of the socket seems questionable. Based on these considerations, a novel, simplified technique, namely, the Biologically-oriented Alveolar Ridge Preservation (BARP) for ARP that restricts socket grafting to the coronal portion of the socket was presented .

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old or more.
* Patients with good oral hygiene, defined as a full-mouth plaque score ≤25% (O'Leary et al., 1972).
* Patients who need alveolar ridge preservation after tooth extraction at one or two sites in the aesthetic zone (incisor, cuspid, or premolar area in the maxilla or mandible) with >50% buccal bone present following tooth extraction (Eeckhout et al., 2022) .
* One or two neighboring teeth.
* Compliant patients who will sign an informed consent and agree to the follow up period.

Exclusion Criteria:

* • Uncontrolled systemic disease

  * Past or current smoking
  * Untreated or unstable periodontitis
  * Untreated caries lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2023-01-05 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Horizontal radiographic changes in bone dimensions | 4 months
  Horizontal measurements will be performed perpendicular and parallel to the tooth axis, respectively. The level of the palatal bone crest preoperatively will be used as a reference line (level 0). The horizontal dimension of the alveolar process will be registered at 1, 3, and 5 mm apical to this reference line (level 1, 3, and 5). After performing all measurements on the CBCT (T1), the software switched to the superimposed image (T4) so that the measurements could be performed while using the same reference levels. Finally, changes in bone dimensions will be calculated by subtracting bone dimensions at T4 from that at T1.

SECONDARY OUTCOMES:
Vertical radiographic changes in bone dimensions | 4 months
  Vertical measurement will be performed by measuring the height of buccal (B) and palatal (p) bone plates from the apical end of the socket to the coronal level of the socket.
Changes of soft tissue height at the buccal , lingual & central aspects of the site. | 4 months
  Since soft tissues will be separated from hard tissues by using lip retractors and a backward position of the tongue, soft tissue height could be assessed on CBCT images. Changes in soft tissue height will be calculated by subtracting soft tissue height at T4 from that at T1

CONTACTS AND LOCATIONS:
Overall Officials: nevein mohmmeda algammal, master, Principal Investigator — phd candidate (assistant lecturer)
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
name: nevein mohammed osama algammal email : nevein.osama@dentistry.cu.edu.eg
Supporting Information: Study Protocol
Time Frame: after completion of the study